CLINICAL TRIAL: NCT05812378
Title: Respiratory Monitoring System Safety and Performance Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RTM Vital Signs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-001
Record Dates: First submitted 2023-04-02; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Function Test; Tidal Volume; Respiratory Rate; Ventilators; Breathing Sounds
Keywords: Minute Ventilation
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

SUMMARY:
The goal of this observational study is collect data to evaluate the efficacy of the RMS system in monitoring, recording, and presenting respiratory function data to the user in participants scheduled for pulmonary function testing (PFT).

Participants will complete:

* 60 episodes of data collection with a decreased tidal volume
* 30 episodes of data collection with an increased tidal volume
* 80 episodes with normal tidal volume breathing

The TSS will continuously transmit sound data to an adjacent personal computer (PC) via Bluetooth Low-Energy (BLE). TSS trachea sound data will be recorded on the PC and then transmitted via a secure wireless network to an RTM cloud account that is HIPPA compliant.

Reference breathing data will be simultaneously recorded using an FDA approved hospital ventilator (Hamilton Medical, HAMILTON-C1) with a calibrated pneumotach, capnometer, and a tight-fitting face mask. This system accurately measures and records a spontaneously breathing patient's RR, TV, MV, and end-tidal carbon dioxide concentration.

DETAILED DESCRIPTION:
Observational single-center data will be captured on up to 50 patients scheduled for pulmonary function testing (PFT) at Thomas Jefferson University Hospital's (TJUH) outpatient PFT facility. Plan is to record a complete data set from 30 patients. Breathing data for this study will be collected in the PFT facility by research personnel approximately 1 hour before or after the scheduled PFT test. Study personnel will adhere the TSS to the skin over the proximal trachea (midline above the sternal notch). The patient's neck will be examined prior to TSS attachment.

The TSS will continuously transmit sound data to an adjacent personal computer (PC) via Bluetooth Low-Energy (BLE). TSS trachea sound data will be recorded on the PC and then transmitted via a secure TJUH wireless network to an RTM cloud account that is HIPPA compliant.

Reference breathing data will be simultaneously recorded using an FDA approved hospital ventilator (Hamilton Medical, HAMILTON-C1) with a calibrated pneumotach, capnometer, and a tight-fitting face mask. This FDA approved system accurately measures and records a spontaneously breathing patient's RR, TV, MV, and end-tidal carbon dioxide concentration.

Study subjects will breathe through the HAMILTON ventilator's face mask, , capnometer, and pneumotach over a range of RR, TV, and MV with the data recorded on a computer. Each study subject will breathe with a normal RR, TV, and MV for approximately 5 minutes. Each subject will then breathe with a normal RR and a decreased tidal volume for approximately 60 to 80 seconds episode (shallow breathing), followed by a rest period (normal breathing). Each subject will then breathe with a normal RR and an increased tidal volume for approximately 60 to 80 seconds episode (deep breathing), followed by a rest period (normal breathing). This series of breathing will take approximately 7.5 minutes to record. Each subject will complete a second series of breathing using the identical methods. Study subjects will observe a computer screen that displays breath- by-breath tidal volume to help them maintain their tidal volume in the desired range during each recording.

Plan is to record and analyze approximately 280 breaths per study subject and 8,400 breaths from the 30 study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to ≤ 80 years
* Subject has no active signs/symptoms of a respiratory infection, severe asthma, severe bronchitis, severe emphysema, or unstable cardiovascular disease at the time of data collection
* Body Mass Index between 18 to 38
* Subject willing and able to comply with the study procedures
* Subject understands the English language, understands the risks, benefits, and alternatives to this research study, and is willing and able to give written informed consent

Exclusion Criteria:

* Subject has an active respiratory infection, unstable cardiovascular disease, severe asthma, severe bronchitis, or severe emphysema at the time of study
* Recent COVID illness (must be symptom free for > 10 days or recent COVID exposure within last 10 days
* History of skin sensitivity to the sensor, adhesive, or face mask materials
* Active inflammation or infection of the skin at the site of TSS attachment
* Subject is pregnant or breastfeeding
* Current participation in another industry sponsored drug or device study
* Patient has a history of anxiety or claustrophobia related to wearing a face mask
* Age < 21 or > 80 years old
* BMI < 18 or > 38

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approximately an equal number of male/female subjects will be studied. Approximately an equal number of subjects will be in the 21 to 40 age range, the 41 to 60 age range, and the > 60 age range. Outpatients scheduled for testing at the PFT Laboratory facility at Thomas Jefferson University Hospital will be recruited for study. Breathing data will be collected by study personnel approximately one hour before or after the scheduled PFT. All patients who meet required inclusion and exclusion criteria are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-12-09 (Estimated); Study Completion 2023-12-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of RMS of the RMS system in monitoring, recording, and presenting respiratory function data to the user | 20 minutes
  The RMS measures respiratory rate, approximate/relative tidal volume, and approximate/relative minute ventilation when compared to measurements made with the HAMILTON ventilator pneumotach device
Mean Measurement Accuracy Error for Respiratory Rate | 20 minutes
  Mean measurement accuracy error for RR across all subjects shall be ≤ 5 % (±1 breath/minute) compared to the pneumotach
Mean Measurement Accuracy Error for Tidal Volume | 20 minutes
  Mean measurement accuracy error for TV across all subjects shall be ≤15% compared to the pneumotach
Mean measurement accuracy error for Minute Ventilation | 20 minutes
  Mean measurement accuracy error for MV across all subjects shall be ≤15% compared to the pneumotach
Mean measurement bias for Respiratory Rate | 20 minutes
  Mean measurement bias (RMS-pneumotach) for RR shall be < 2% (95% limits of agreement ±1.96 SD)
Mean measurement bias for Tidal Volume | 20 minutes
  Mean measurement bias (RMS-pneumotach) for TV shall be < 5% (95% limits of agreement ±1.96 SD)
Mean measurement bias for Minute Ventilation | 20 minutes
  Mean measurement bias (RMS-pneumotach) for MV shall be < 5% (95% limits of agreement ±1.96 SD)
Tidal volume trend | 20 minutes
  Tidal volume trend > 0.95 (r² correlation to pneumotach)
Mean measurement accuracy error for number of seconds since last breath | 20 minutes
  Mean measurement accuracy error for number of seconds since last breath across all subjects shall be ≤ 5 % (± 2 seconds) compared to the pneumotach

CONTACTS AND LOCATIONS:
Overall Officials: Marc Torjman, PhD, Principal Investigator — Thomas Jefferson University and Hospitals Department of Anesthesiology and Perioperative Medicine
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States